CLINICAL TRIAL: NCT03517397
Title: Mobile Contingency Management for Smoking Cessation Among Socioeconomically Disadvantaged Adults
Brief Title: Mobile Contingency Management for Smoking Cessation (R01 Supplement) (PrevailGO)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7210; R01CA197314 (NIH)
Record Dates: First submitted 2018-03-30; First posted 2018-05-07 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Smoking Cessation
Keywords: Smoking Cessation; Socioeconomic Disadvantage; Contingency Management; Financial Incentives; Mobile Health; Biochemical Verification
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile Contingency Management (Experimental)
  Interventions: Behavioral: Mobile Contingency Management

INTERVENTIONS:
Behavioral: Mobile Contingency Management — Participants will be offered 6 counseling sessions, nicotine replacement therapy, and a smartphone app that remotely verifies participant identity and smoking abstinence and automatically credits a gift card account for evidence of smoking abstinence.

SUMMARY:
Smoking prevalence rates are disproportionately high among individuals living below the poverty threshold, those living in rural areas, and Oklahomans. Nearly 1.3 million Oklahomans live in rural areas and the prevalence of poverty is elevated relative to the U.S. Our preliminary work has indicated that offering small escalating financial incentives for smoking abstinence (i.e., Contingency Management [CM]) dramatically increases short-term cessation rates among socioeconomically disadvantaged smokers when incentives are included as an adjunct to clinic-based smoking cessation treatment. However, other approaches are needed for socioeconomically disadvantaged individuals who are unable to attend clinic visits due to rural residence or other limitations. Internet and mobile phone-based CM approaches have been developed to reduce or eliminate the need for in-person visits. The goal of the current project is to improve upon existing mobile CM approaches by fully automating the process to make financial incentives interventions for smoking cessation feasible and accessible to individuals across the state. The aims of the proposed project are to 1) develop a fully automated, mobile phone-based CM approach to remotely verify smoking abstinence, confirm participant identity, and deliver financial incentives for smoking cessation, and 2) evaluate the feasibility and preliminary effectiveness of using fully automated mobile CM as an adjunct to telephone counseling and nicotine replacement therapy among 20 socioeconomically disadvantaged adults. The current project extends the scope of the parent study by increasing the reach of the CM approach to socioeconomically disadvantaged individuals who may be unable to attend in-person visits.

DETAILED DESCRIPTION:
Tobacco Cessation Treatment. Participants referred to the Tobacco Treatment Research Program (TTRP) for smoking cessation treatment who are interested and eligible for the current study will be offered weekly telephone counseling/support sessions led by a staff counselor. Six unique sessions covering the following topics will be offered: 1) quit planning 2) the impact of tobacco on health/benefits of quitting, 2) stress management strategies, 3) making positive lifestyle changes, 4) developing coping skills, and 5) relapse prevention. The counselor will check in with participants each week about the difficulties and successes they have experienced, and plan for any challenging situations that are anticipated. Advice and support will be provided as needed. A two-week supply of nicotine replacement therapy (patches and gum) will be offered during the first session for medically eligible participants. Additional patches and gum will be mailed out for participants who wish to continue using pharmacotherapy (for up to 12 weeks).

Financial Incentives. Participants will be provided with a smartphone that has the PrevailGO EMA app preloaded, as well as a Smokerlyzer iCO monitor. Participants will be randomly prompted 4 times daily during waking hours to complete smartphone-based EMAs. During random prompts, participants who self-report abstinence will be asked to provide a CO breath sample on 5 randomly selected days out of the week. Participants will be prompted to provide a CO breath sample at the last random assessment of the day, Participants will be reminded 2 additional times on the same day during their normal waking hours to provide a CO breath sample if they miss the initial assessment. A gift card credit may be earned following a self-report of abstinence during the past 24 hours combined with a breath CO sample of ≤ 6 ppm.

Recruitment/Screening (Visit 1, Part 1; Screening). Individuals who are referred to the TTRP for smoking cessation treatment and report that they are uninsured or receiving Medicaid benefits will be sent an informational handout with their TTRP information packet (prior to their first visit). Participants will be reminded of all future in-person appointments via telephone, mail, email, and/or text. Additionally, research staff may attempt to collect smoking cessation status with each reminder. Participants with transportation difficulties living in the Oklahoma City metro area may be scheduled for pick-up and drop-off for key visits with SendaRide through their secure dashboard. At the first visit, study staff will inquire about their interest in finding out more about the study. Study staff will review the consent form with interested participants, and they will be screened for eligibility on-site in a private room in the clinic. Participant eligibility for the current study will not influence eligibility for the TTRP. The Rapid Estimate of Adult Literacy in Medicine (REALM; see Appendix A) will be administered to ensure that all participants are able to read at ≥ sixth grade level (i.e., required to complete EMA and self-report questionnaires). Expired carbon monoxide (CO) will be measured and participants will be questioned about their 1) insurance status 2) age, 3) current level of smoking, 4) willingness to quit smoking, 5) willingness/ability to complete 6 weekly counseling sessions (including the first visit), 6) pregnancy/breastfeeding status, 7) computer/internet access, and 8) contraindications for nicotine replacement therapy. Expired CO will be measured. Eligible participants may complete the assessment portion of the visit.

Pre-Quit (Visit 1, Part 2; Assessment). Participants will complete self-report questionnaires on a laptop computer; weight and height will be measured in a private room to ensure confidentiality. Visit 1 will be 1 of 2 in-person visits. Participants will be provided with an Android smartphone and a Smokerlyzer iCO breathe monitor. They will be instructed regarding the use of the phone (participants may make personal calls), the EMA procedures, and use of the portable CO monitor. Participants will receive 4 random prompts and 1 daily diary prompt (in the morning) during the normal waking hours each day for five consecutive weeks. Participants will be instructed to quit smoking at bedtime or 10:00 pm (whichever occurs first) 7 days after enrollment.

Quit Day. Participants will remotely complete web-based self-report questionnaires and provide a smartphone-based CO measurement.

One Week Post-Quit. Participants will remotely complete web-based self-report questionnaires and provide a smartphone-based CO measurement.

Two Weeks Post-Quit. Participants will remotely complete web-based self-report questionnaires and provide a smartphone-based CO measurement.

Three Weeks Post-Quit. Participants will remotely complete web-based self-report questionnaires and provide a smartphone-based CO measurement.

Four Weeks Post-Quit. Participants will remotely complete web-based self-report questionnaires and provide a smartphone-based CO measurement.

Eight Weeks Post-Quit. Participants will remotely complete web-based self-report questionnaires and provide a smartphone-based CO measurement.

Twelve Weeks Post-Quit. Participants will return to the TTRP and complete self-report questionnaires on a tablet or laptop computer and provide a CO measurement.

ELIGIBILITY:
Inclusion Criteria:

* currently uninsured or receiving Medicaid benefits
* earn a score ≥ 4 on the REALM indicating > 6th grade English literacy level
* willing to quit smoking 7 days from their first visit
* 18-64 years of age
* expired CO level ≥ 8 ppm suggestive of current smoking
* currently smoking ≥ 5 cigarettes per day
* own or have access to a computer (to remotely complete study questionnaires).

Exclusion Criteria:

* pregnant or breastfeeding
* have uncontrolled hypertension
* had a myocardial infarction within the past two weeks
* have an allergy to adhesive tape
* are unwilling to use nicotine replacement therapy.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Biochemically-verified smoking cessation | 12 weeks post-quit date
  Self-reported abstinence over the past 7 days in conjunction with a carbon monoxide value < 6 ppm
Treatment Participants | 5 weeks post-enrollment
  Treatment sessions completed (1-6)
Follow-Up Completion Rate | 12 weeks post-quit date
  The number of people who provide self-reports of smoking status and biochemical verification of smoking cessation.

SECONDARY OUTCOMES:
Device Loss | 13 weeks post-enrollment
  The total number of phones and iCO monitors lost.
Completion of Ecological Momentary Assessment | 5 weeks post-enrollment
  Percentage of ecological momentary assessments completed

CONTACTS AND LOCATIONS:
Overall Officials: Darla E. Kendzor, PhD, Principal Investigator — The University of Oklahoma Health Sciences Center
Locations (1):
- The University of Oklahoma Health Sciences Center, Tobacco Treatment Research Program, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kendzor DE, Businelle MS, Waring JJC, Mathews AJ, Geller DW, Barton JM, Alexander AC, Hebert ET, Ra CK, Vidrine DJ. Automated Mobile Delivery of Financial Incentives for Smoking Cessation Among Socioeconomically Disadvantaged Adults: Feasibility Study. JMIR Mhealth Uhealth. 2020 Apr 15;8(4):e15960. doi: 10.2196/15960. PMID 32293568